CLINICAL TRIAL: NCT03374748
Title: Examination of Varying Statistical Methods to Determine Meal Patterns Using Data From the National Adult Nutrition Survey (NANS) Ireland.
Brief Title: Examination of Meal Patterns in National Adult Nutrition Survey (NANS), Ireland
Status: Completed | Type: Observational
Sponsor: University College Dublin (Other)
Collaborators: University College Cork (Other)
Responsible Party: Sponsor
Other Study IDs: NANS_MealPatterns_UCD
Record Dates: First submitted 2017-12-06; First posted 2017-12-15 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Food Consumption Database Analysis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and Urine Collection and Analysis - Participants were asked to provide a blood sample, fasting where possible, and a first void morning urine sample. The blood tubes collected were: 3 x serum tubes (total 26ml); 2 x EDTA tubes (total 13ml); 1 x lithium heparin tube (6ml). A 50ml first void urine sample was also collected. Blood and urine samples were collected for the analysis of a number of markers of nutritional status and metabolic health.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: N/A - observational study — N/A - observational study

SUMMARY:
This study is a secondary analysis of the dietary, phenotypic and demographic data collected within the National Adult Nutrition Survey (NANS), Ireland, to determine meal patterns using a variety of statistical methods.

DETAILED DESCRIPTION:
The study described here applies a variety of statistical methods to develop strategies to determine meal based dietary patterns within nationally representative food consumption databases. The work will apply methods such as Principal component analysis, latent class analysis, basket set analysis, topic models and others to explore methods to accurately identify meal based dietary patterns for use in personalised nutrition.

The work will initially focus on National Food Consumption Data collected within Ireland, specifically using the National Adult Nutrition Survey (NANS), with details of data collection fully outlined below.

Within NANS dietary, demographic and phenotypic data was collected from a Nationally representative sample within Ireland from 2008-10. The fieldwork phase was carried out between October 2008 and April 2010. Adults aged 18-90 years (740 males, 760 females) were recruited in the Republic of Ireland. Eligible respondents were adults aged 18 years and over who were free-living and who were not pregnant or breast feeding. A sample of adults was randomly selected from a database of names and addresses held by Data Ireland (An Post). An introductory letter and information leaflet were posted to each person selected from the database. A researcher called to potential respondents" homes to introduce the survey and invite participation. If the individual agreed to participate, a consent form was signed and the survey commenced. If the person was not at home, the researcher called on three more occasions on different days and at different times, before deeming them ineligible. For groups that were not highly represented in the database, particularly 18-35 year olds, a second level of recruitment was introduced. A second database of names and addresses was compiled through referrals from respondents and participation was invited for those that were contactable.

Food intake data collection - A four-day food diary was used to collect food and beverage intake data. The researcher made three visits to the respondent during the four-day period: a training visit to demonstrate how to keep the food diary and how to use the weighing scales; a second visit 24-36 hours into the recording period to review the diary, check for completeness and clarify details regarding specific food descriptors and quantities; and a final visit one or two days after the recording period to check the last days and to collect the diary. Respondents were asked to record detailed information regarding the amount and types of all foods, beverages and nutritional supplements consumed over the recording period and where applicable, the cooking methods used, brand names of the foods consumed and details of recipes. Data were also collected on the time of each eating or drinking occasion, the respondent's definition of each eating or drinking occasion (e.g. morning snack, lunch) and the location of the preparation of the meal or snack consumed.

Food quantification and coding - A quantification protocol that had been established by the IUNA (Irish Universities Nutrition Alliance) for the North/South Ireland Food Consumption Survey (NSIFCS) (Harrington et al., 2001) was updated for the NANS. It is summarised as follows: (1) Weighed by respondent/manufacturer weights) - A portable food scales (Tanita, Japan) was given to each respondent. The researcher gave detailed instructions (including a demonstration) as to how to use the food scales during the training session. This method was use to quantify 46% of foods and drinks consumed. A further 10% of weights were derived from manufacturer's weights. To facilitate collection of such data, researchers asked respondents to collect all packaging of food and beverages consumed in a storage bag provided. (2) Food Atlas - A photographic food atlas (Nelson et al., 1997) was used to quantify 16% of foods and beverages consumed. (3) IUNA Weights - Average portion weights that had been ascertained for certain foods by the IUNA survey team were used. This method was used to quantify 4% of foods and beverages consumed. (4) Food Portion Sizes - "Food Portion Sizes" (Ministry of Agriculture, Fisheries and Food, 1997) was used to quantify 11% of foods and beverages consumed. (5) Household Measures - Measures such as teaspoon, tablespoon, pint etc. were used to quantify 11% of foods and beverages consumed. (6) Estimated - Food quantities were defined as estimated if the researcher made an estimate of the amount likely to have been consumed based on their knowledge of the respondent's general eating habits as observed during the recording period. This method was used to quantify 2% of foods and beverages consumed. Nutrient composition of foods and estimation of nutrient intake - Food intake data were analysed using WISP© (Tinuviel Software, Anglesey, UK). WISP© uses data from McCance and Widdowson's The Composition of Foods, sixth (Food Standards Agency, 2002) and fifth (Holland et al., 1995) editions plus all nine supplemental volumes (Holland et al., 1988; Holland et al., 1989; Holland et al., 1991; Holland et al., 1992; Holland et al., 1993; Chan et al., 1994; Chan et al., 1995; Chan et al., 1996; Holland et al., 1996) to generate nutrient intake data. During the NANS, modifications were made to the food composition database to include recipes of composite dishes, nutritional supplements, generic Irish foods that were commonly consumed and new foods on the market. All previous modifications to the food composition database were also checked and updated from current manufacturers" information as necessary. The above modifications and additions comprise "The Irish Food Composition Database" (Black et al., 2011).

Questionnaires - Four questionnaires were completed by the adults in the NANS. These included: Health and Lifestyle Questionnaire: This questionnaire collected information on the respondent's socio-demographics, education levels, attitudes to their own diet and weight, sun exposure and supplement usage. Information on smoking status and alcohol intake was also collected in this questionnaire. In the case of married/cohabiting couples, the higher social class and education level was assigned to the respondent.

Physical Activity: Respondents completed a validated physical activity questionnaire (Epic Physical Activity Questionnaire (EPAQ2)) (Wareham et al. 2002) to assess customary levels of physical activity. The questionnaire consisted of three sections: activity at home, work and recreation.

Food Choice Questionnaire: This questionnaire was designed to find out information on food choice and the factors that can influence it, fear of eating new or unfamiliar foods and the respondent's own opinion of their food preparation skills. Evaluation Questionnaire: The researcher administered this questionnaire at the final visit to identify whether the respondent's eating habits or physical activity patterns had been usual during the survey week. Medication usage was also recorded here. Coded questionnaires were entered into the customised Q-Builder software package (Tinuviel Software, Anglesey, UK). A dual data entry method was used to enter questionnaires to ensure correct data entry.

Anthropometry - Anthropometric measurements were taken by the researcher in the respondents" homes. Weight, height, waist and hip circumference and measures of body composition were recorded. Height was measured to the nearest 0.1cm using the Leicester portable height measure (Chasmores Ltd, UK) with the respondent's head positioned in the Frankfurt Plane. Waist circumference was measured in duplicate using a non-stretch tape measure and taken at the naked site where possible. Waist circumference was measured at the midpoint to the nearest 0.1cm between the iliac crest (top of hip) and the bottom of the rib cage (10th rib). Hip circumference was measured in duplicate to the nearest 0.1cm using a non-stretch tape measure. This measurement was taken over light clothing at the widest part of the buttocks at the level of the greater trochanter (bony prominence of the thigh bone). Weight and body composition were measured in duplicate using a Tanita body composition analyzer BC-420MA (Tanita Ltd, GB) to the nearest 0.1kg. Respondents were weighed after having voided, wearing light clothing and without shoes. Defining overweight and obesity in adults Body Mass Index (BMI) was used to indirectly assess adiposity and was calculated as weight (kg) divided by height squared (m2). The World Health Organisation (WHO) BMI cut-off points were used to estimate levels of underweight (<18.5kg/m2), normal weight (18.5-24.9kg/m2), overweight (25.0-29.9kg/m2) and obese (≥30 kg/m2).

Blood Pressure - Blood pressure was measured in triplicate from the right arm where possible, leaving five minutes between each measurement. The measurement was taken with the respondent sitting on a well-supported chair, with feet placed firmly on the floor. Prior to the measurement, respondents were asked to sit quietly without talking or laughing for at least five minutes. Respondents were asked to remove tight clothing from their upper arm and to rest their arm such that the antecubital fossa (triangular cavity of the elbow joint) was at the level of the heart, palm facing upwards. Measurements were taken in accordance with the manufacturer's instructions for the OMRON M6 Comfort blood pressure monitor, with fieldworkers having received training in taking the measurement prior to fieldwork. Respondents were asked whether they had had anything to eat or drink (besides water) or whether they had smoked in the 30 minutes prior to the measurement. This information was recorded by the fieldworker. Respondents were informed of blood pressure readings that consistently fell outside of the normal ranges and advised to visit their health nurse or general practitioner for another reading.

Blood and Urine Collection and Analysis - Participants were asked to provide a blood sample, fasting where possible, and a first void morning urine sample. The samples were collected by a qualified nurse at designated centres within the survey area or in the respondent's home if the respondent could not travel. In total, five tubes (45mls) of blood were collected from respondents and where appropriate, inverted gently to ensure thorough mixing with anti-coagulant. Of these, four were kept chilled and transported to the lab for further processing and storage, while the fifth was kept at room temperature for full blood count analysis. The blood tubes collected were: 3 x serum tubes (total 26ml); 2 x ethylenediaminetetraacetic acid (EDTA) tubes (total 13ml); 1 x lithium heparin tube (6ml). A 50ml first void urine sample was also collected. Respondents were provided with a sterile collection tube to collect the urine sample on the final survey visit. They were also provided with an ice pack and asked to keep the sample chilled until they met with the nurse. Samples were kept on ice during transport to the lab for further processing. A blood collection form was completed in which the following was recorded: date and time of blood collection, whether the respondent was fasting or not and any irregularities during blood collection. Written consent to take a blood and urine sample was obtained along with consent for the survey at the initial visit. Blood and urine samples were collected for the analysis of a number of markers of nutritional status and metabolic health. In line with good ethical practice, all samples were anonymised prior to analysis.

Physical activity and accelerometer - A triaxial accelerometer (Actigraph GT1M, ActiGraph, LLC) was worn for the four days of the survey period. It was worn on the waist and reported acceleration using a proprietary unit - "counts". An accelerometer diary was also used to track activities that are poorly recorded by accelerometers such as cycling and swimming and to record when the accelerometer was removed e.g. for sleeping/showering.

ELIGIBILITY:
Inclusion Criteria:

Eligible respondents were adults aged 18 years and over who were free-living

Exclusion Criteria:

Individuals who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The fieldwork phase was carried out between October 2008 and April 2010. Eligible respondents were adults aged 18 years and over who were free-living and who were not pregnant or breast feeding. A sample of adults was randomly selected from a database of names and addresses held by Data Ireland (An Post).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Food intake | 4 days
  Food intake measured using semi weighed food diary

CONTACTS AND LOCATIONS:
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
Access to the primary data is available through application to www.iuna.net or the PI Prof Albert Flynn University College Dublin.

REFERENCES:
- [Derived] Jarrett H, McNulty H, Hughes CF, Pentieva K, Strain JJ, McCann A, McAnena L, Cunningham C, Molloy AM, Flynn A, Hopkins SM, Horigan G, O'Connor C, Walton J, McNulty BA, Gibney MJ, Lamers Y, Ward M. Vitamin B-6 and riboflavin, their metabolic interaction, and relationship with MTHFR genotype in adults aged 18-102 years. Am J Clin Nutr. 2022 Dec 19;116(6):1767-1778. doi: 10.1093/ajcn/nqac240. PMID 36264281